CLINICAL TRIAL: NCT04812080
Title: EXPLORER PET/CT: Evaluation of Healthy Individuals From Racial/Ethnic Minority Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1714742
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Results first posted 2023-02-15 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers From Racial/Ethnic Minority Populations

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EXPLORER PET/CT Imaging (Experimental): Study participants will be injected with 10 +/- 2 mCi of 18F-FDG using and IV line and a 60 minute PET scan will begin on EXPLORER. Prior to the PET scan, an ultra-low-dose CT scan (less than 1 minute ) will be acquired for attenuation correction purposes only. Ninety (90) minutes after being injected with FDG, participants will have another ultra-low dose CT scan (less than 1 minute) which will be acquired for attenuation correction purposes only. This will be followed by a 20 minute PET scan on EXPLORER. One-hundred and twenty (120) minutes after being injected with FDG, participants will be positioned supine on the scanner table for the last time. At this time, a low dose CT scan (less than 1 minute) will be acquired once again for attenuation correction purposes. This will be followed by one last 20 minute PET scan on EXPLORER. The IV line will be removed after completion of the study.
  Interventions: Device: EXPLORER PET/CT

INTERVENTIONS:
Device: EXPLORER PET/CT — FDG PET Scans on the total body EXPLORER PET/CT scanner

SUMMARY:
The objective of this pilot study is to collect preliminary data using total body scans on a new, first of its kind, FDA 510k-cleared positron emission tomography/computed tomography (PET/CT) scanner, called EXPLORER. The study will aim to recruit healthy individuals from racial/ethnic minority populations.

DETAILED DESCRIPTION:
The aim of this pilot study is to increase the number of healthy individuals from racial/ethnic minority populations. This will advance research being conducted at EMIC by providing "controls" or comparisons to differentiate between images from patients with cancer versus healthy people of the same racial/ethnic ancestry. In addition, blood samples from participants to this study will be utilized for quantitative, genetics-based estimates of ancestry (e.g., African, Chinese, Colombian, Western European, Mexican, Vietnamese, etc.), which is especially valuable in the case of admixed individuals.

ELIGIBILITY:
Inclusion criteria:

* Men and women, 18 years of age or older
* Member of a Federally recognized racial/ethnic minority population, e.g., African American or Black; Hispanic or Latino; Asian American; Native Hawaiian or Other Pacific Islander; Native American or Alaska Native
* Willing and able to fast for at least 6 hours before and for the duration of the scan
* Willing to provide urine samples throughout scan visit
* Willing to provide blood samples for ancestry analysis
* Willing and able to lay motionless in a supine position for up to 60 minutes and for up to 20 minutes at two separate timepoints
* Willing and able to give informed consent, personal contact information (phone number, email and postal address), insurance information, and primary care physician contact

Exclusion criteria:

* No Primary Care Physician
* No health insurance
* Body weight more than 240 kg (529 pounds)
* Any known concomitant acute infection (including upper respiratory infection, genitourinary infections, etc.)
* History of metastatic or newly (last 5 years) diagnosed locally invasive cancer
* Chemotherapy in the last 5 years
* Radiation therapy in the last 3 years
* Major surgery within the last 6 months
* Pregnancy or breast-feeding
* Diabetes
* Fasting blood glucose level > 200 mg/dL before administration of fluorodeoxyglucose (FDG)
* Prisoners
* Self-reported history of dysphoria or anxiety in closed spaces

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moon Chen, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EXPLORER PET/CT Imaging
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | EXPLORER PET/CT Imaging
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 51.52 [27 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Standardized Uptake Value (SUV) in gm/ml Reported as Mean and Standard Deviation
Description: To collect preliminary data about total body FDG perfusion and early biodistribution in a cohort of racial/ethnic minority volunteers as measured by standardized uptake value (SUV) in gm/ml reported as Mean and Standard Deviation. The SUV is the ratio of the image-derived radioactivity concentration and the whole body concentration of the infected radioactivity.
Time Frame: 3 hours
Population: All the participants completed their scheduled scans at three timepoints: dynamic scan for 60 minutes, two scans at 90- and 120-minutes post-injection, for 20-minutes each.
Measure: Mean (Standard Deviation); unit: gm/ml
Arm/Group | EXPLORER PET/CT Imaging
Number analyzed (Participants) | 20
gm/ml
  Brain @ 40 minutes | 7.293 (1.678)
  Brain @ 90 minutes | 5.157 (1.323)
  Brain @ 120 minutes | 4.429 (1.141)
  Aorta @ 40 minutes | 2.357 (0.208)
  Aorta @ 90 minutes | 1.039 (0.123)
  Aorta @ 120 minutes | 0.794 (0.089)
  Liver @ 40 minutes | 2.639 (0.285)
  Liver @ 90 minutes | 1.215 (0.156)
  Liver @ 120 minutes | 0.966 (0.109)
  Spleen @ 40 minutes | 2.029 (0.254)
  Spleen @ 90 minutes | 1.019 (0.130)
  Spleen @ 120 minutes | 0.846 (0.130)
  Vertebrae @ 40 minutes | 1.380 (0.186)
  Vertebrae @ 90 minutes | 0.839 (0.137)
  Vertebrae @ 120 minutes | 0.712 (0.125)
  Skeletal muscle @ 40 minutes | 0.768 (0.068)
  Skeletal muscle @ 90 minutes | 0.425 (0.052)
  Skeletal muscle @ 120 minutes | 0.353 (0.049)
  Subcutaneous fat @ 40 minutes | 0.451 (0.078)
  Subcutaneous fat @ 90 minutes | 0.207 (0.037)
  Subcutaneous fat @ 120 minutes | 0.155 (0.027)

2. Primary Outcome: Count of Participants With Confirmed Ancestry Informative Markers
Description: Participants' self-reported racial/ethnic identity and ancestral origin confirmation with Ancestry Informative Markers (AIMS) analysis
Time Frame: 15 minutes
Measure: Count of Participants; unit: Participants
Groups:
- EXPLORER PET/CT Ancestry Informative Markers: Genetic Ancestry Informative Markers compared to self report from participants
Arm/Group | EXPLORER PET/CT Ancestry Informative Markers
Number analyzed (Participants) | 20
Participants | 20

ADVERSE EVENTS:
Time Frame: AEs were collected during the study protocol activity of the one appointment for approximately 3 hours at which time the subject was off study.
Arm/Group | EXPLORER PET/CT Imaging
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT04812080/Prot_SAP_ICF_001.pdf